CLINICAL TRIAL: NCT01800149
Title: Healing of Post-extraction Sites Using Bovine-bone Mineral: a CBCT and Histologic Randomized Controlled Clinical Study
Brief Title: Healing of Post-ext Sites Using Bovine Bone Mineral: a CBCT and Histologic RCCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Proed, Torino, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01.2013.POST-EXT.PROED
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Loss of Teeth Due to Extraction; Edentulous Alveolar Ridge
Keywords: Tooth extraction; Ridge Preservation; Ridge Augmentation; Guided Bone Regeneration
MeSH Terms: interventions — Alveolar Ridge Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BBM+collagen (Active Comparator): Ridge Augmentation After tooth extraction, edentulous sockets will be filled with BioOss Collagen and covered with Bio-Gide
  Interventions: Procedure: Ridge Augmentation
- BBM granules (Active Comparator): Ridge Augmentation After tooth extraction, edentulous sockets will be filled with Bio-Oss Granules, 0-25-1 mm, and covered with Bio-Gide
  Interventions: Procedure: Ridge Augmentation

INTERVENTIONS:
Procedure: Ridge Augmentation — After tooth extraction, the sockets will be filled with bovine bone mineral and covered with a porcine collagen membrane

SUMMARY:
Aim of the present investigation will be to evaluate the role of a bovine-bone mineral and a collagen membrane as ridge augmentation procedure following tooth extraction. 20 consecutive adult patients, requiring tooth extraction in the frontal area of the upper and lower arch maxilla (from second premolar to second premolar), will be enrolled into the study.

After tooth extraction, sockets will be randomized and divided into two groups: in Group A the socket will be grafted with Bio-Oss Collagen , in Group B the sockets will be grafted with BioOss granules (small granules). The graft will be covered with porcine collagen membrane (BioGide). Then, the flap will be sutured.

MEASUREMENTS:

The end of the study will be fixed at the 6 months evaluation after tooth extraction. Impression will be taken before tooth extraction and after 6 months in order to create cast models. On the cast models, using reference PVC (polyvinylchloride) guides, the horizontal dimension of the soft tissues will be measured. One measurement per tooth will be recorded, at T0 (before extraction) and T2 (after 6 months).

A 3D radiological image, using the CBCT technique, will be obtained at the end of the surgical stage T1 (extraction + bone graft) and after 6 months of healing. Superimposition will be performed in order to measure hard tissue remodelling.

After six months (T6), a a biopsy specimen will be also harvested for that augmented extractions sockets on which an implant installation has been previously planned.

DETAILED DESCRIPTION:
Both animal and human studies have clearly demonstrated that the healing of post extraction sites usually results in pronounced alveolar ridge resorption, that mostly stabilized after 4 to 6 months. The marked tri-dimensional alterations of the ridge volume may jeopardize patients' aesthetics and create anatomical difficulties for further implant placement.

Aim of the present investigation will be to evaluate the role of a bovine-bone mineral and a collagen membrane as ridge augmentation procedure (intended as "increase of the ridge volume beyond the skeletal envelope existing at the time of extraction") following tooth extraction. Furthermore, the authors aim to evaluate as the collagen membrane acts when used for "open-healing".

20 consecutive adult patients, requiring tooth extraction in the frontal area of the upper and lower arch maxilla (from second premolar to second premolar), will be enrolled into the study.

After local anesthesia, a buccal full thickness flap will be elevated, and then the hopeless teeth will be gently extracted. All granulation tissue will be removed from the alveolus, that will be rinsed with saline. At this time the post-extraction sockets will be randomized and divided into two groups: in Group A the socket will be grafted with Bio-Oss Collagen , in Group B the sockets will be grafted with BioOss granules (small granules) using the Bio-Oss Pen device.

The graft will be covered with porcine collagen membrane (BioGide). Then, the flap will be sutured. The sutures (single sutures) will involve only the interdental gingival tissue, and no attempt will be done to reach a complete soft tissue closure of the sockets: in the alveolus area BioGide will be mostly left exposed, intended as "open healing" for second intention wound healing.

The patient swill assume antibiotics per 6 days (Amoxicillin + Clavulanate 1gr), and will rinse with Digluconate Chlorhexidine 0.20% per 14 days. At day 14 the sutures will be removed. If, at this moment, the gingiva over the graft will not be completely closed, the patient will use Digluconate Chlorhexidine 0.20% until the secondary closure will be completed.

MEASUREMENTS:

The end of the study will be fixed at the 6 months evaluation after tooth extraction (corresponding to the planned time for implant installation).

Impression will be taken before tooth extraction and after 6 months in order to create cast models. On the cast models, using reference PVC guides, the horizontal dimension of the soft tissues (measured perpendicular to the tangent of the dental arch at the midpoint of the extraction site as the distance between the most prominent points buccally and orally) will be measured. One measurement per tooth will be recorded, at T0 (before extraction) and T2 (after 6 months).

A 3D radiological image, using the CBCT technique, will be obtained at the end of the surgical stage T1 (extraction + bone graft) and after 6 months of healing. Using a diagnostic software, superimposition will be performed in order to measure hard tissue remodelling.

After six months (T6), a a biopsy specimen will be also harvested for that augmented extractions sockets on which an implant installation has been previously planned, with the purpose of an histologic and histomorphometric evaluation (measurement of new bone formation and measurement of remaining BioOss granules). The biopsy will be taken exactly in the area where dental implants will be placed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients with one or more teeth to be extracted, from premolar to premolar

Exclusion Criteria:

* Heavy smokers (more than 10 cig per day)
* Current Pregnant patients
* History of malignancy
* History of radiotherapy or chemiotherapy in the past 5 years
* Long term steroidal or antibiotic therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical horizontal width | 6 months after tooth extraction
  On the cast models, using reference PVC stants, the horizontal dimension of the soft tissues (measured perpendicular to the tangent of the dental arch at the midpoint of the extraction site as the distance between the most prominent points buccally and orally) will be measured.

SECONDARY OUTCOMES:
Radiological horizontal width | 6 months after tooth extraction
  A 3D radiological image, using the CBCT technique, will be obtained at the end of the surgical stage T1 (extraction + bone graft) and after 6 months of healing. Using a diagnostic software, superimposition will be performed in order to measure hard tissue remodelling.

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Cardaropoli, DDS, Study Director — Proed, Torino, Italy
Locations (1):
- PROED, Institute for Professional Education in Dentistry, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: No